CLINICAL TRIAL: NCT06738979
Title: A Multicenter, Randomized, Open, Parallel Controlled Phase III Study Comparing the Efficacy and Safety of Semaglutide Injection and Wegovy® for Weight Management in Obese Subjects
Brief Title: A Clinical Study Comparing Semaglutide Injection and Wegovy® for Weight Management in Obese Subjects
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQF3510-III-02
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — semaglutide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQF3510 (Experimental): TQF3510: The drug treatment cycle was 44 weeks, including a dose escalation period of 16w and a stable dose period of 28w.
  Interventions: Drug: TQF3510 (Semaglutide Injection)
- Wegovy® (Active Comparator): Wegovy® : The drug treatment cycle consisted of a dose escalation period of 16w and a stable dose period of 28w.
  Interventions: Drug: Wegovy®

INTERVENTIONS:
Drug: TQF3510 (Semaglutide Injection) — Semaglutide injection is a long-acting Glucagon-like peptide-1 (GLP-1) receptor agonist.
  Arms: TQF3510
Drug: Wegovy® — Active Comparator
  Arms: Wegovy®

SUMMARY:
This is a multicenter, randomized, open, parallel, positive-controlled clinical study to evaluate the efficacy and safety of Semaglutide injection (TQF3510) developed by Chia Tai Tianqing Pharmaceutical Group Co., Ltd. in obese subjects (BMI≥28 kg/m2).

Equivalence tests were performed for the percentage (%) of weight loss at 44w relative to baseline at the primary endpoint. A meta-analysis was performed based on multiple registration studies of the original drug Wegovy® (semaglutide), and the final equivalence threshold was determined (-4.16%, 4.16%). It was assumed that the sample size ratio of the experimental group and the control group was 1:1, the overall difference between the experimental group and the control group was 0, the standard deviation of the reference original drug was 11%, and the degree of assurance (1-β) was 85%. Double unilateral t test was adopted, and double unilateral α=0.025. The sample size was 326 cases by the Power Analysis & Sample Size (PASS) 2019 Software. Considering the 20% shedding rate, 408 patients were enrolled in this study, 204 in each group.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old, gender is not limited;
* Body mass index (BMI) ≥ 28 kg/m2;
* Self-report at least one unsuccessful diet and weight loss history;
* Patients must give informed consent to this study before the trial and sign the informed consent voluntarily.

Exclusion Criteria:

* Pregnant or lactating women or men or women of childbearing age who had a pregnancy plan during the study period (including a spouse), or who refused to take the contraceptive measures specified in the programme during the study period;
* Have a history of diabetes of any type;
* Patients who had used any hypoglycemic drugs within 90 days before screening;
* Personal or first-degree relatives have a personal or family history of thyroid C-cell tumor or multiple endocrine tumor syndrome type 2;
* Use of any drugs for weight management within 90 days prior to screening;
* Previous or planned weight loss related treatment through surgery or other weight loss means during the study period;
* Have a history of major depression or serious mental illness;
* Mental Health Scale (PHQ-9) score ≥ 15 during screening;
* History of acute pancreatitis within 180 days prior to screening;
* Have a history of chronic pancreatitis or pancreatic surgery;
* Laboratory tests during screening meet any of the following criteria:

  1. Alanine aminotransferase (ALT)> 2.5× upper limit of normal (ULN), aspartate aminotransferase (AST)>2.5 ULN;
  2. Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m2;
  3. calcitonin ≥ 50 ng/L (pg/mL);
  4. Triglyceride (TG) ≥500 mg/dl (5.7mmol/L);
  5. Thyroid stimulating hormone (TSH) >6 mIU/L or <0.4 mIU/L.
* When virological tests at the time of screening show any of the following:

  1. Hepatitis C virus (HCV) antibody positive, and HCV virus titer detection value exceeds the upper limit of normal value;
  2. HBsAg positive and Hepatitis B virus (HBV) DNA test value exceeds the upper limit of normal value;
  3. HIV positive;
  4. Active syphilis: the screening period of treponema pallidum antibody positive and non-Treponema pallidum serum test (RPR or TRUST) positive;
* Uncontrolled or poorly treated hypertension;
* Clinically significant cardiovascular and cerebrovascular disease in the 6 months prior to screening;
* People who are allergic to Semaglutide injection or any component of Wegovy®, or to other GLP-1 receptor agonists, or who have a pre-existing allergic disorder;
* Participated in any other clinical trial within 3 months prior to screening;
* The subject is unable to comply with the treatment plan and diet and exercise plan established by the investigator;
* There are secondary causes affecting body weight;
* There is hypothyroidism at the time of screening that is not controlled with stable drug dosages;
* Have a history of major surgery within 6 months prior to screening;
* A history of drug abuse or alcohol dependence within the 6 months prior to screening;
* History of malignant tumor within 5 years before screening;
* Patients with other diseases that the researchers assessed would affect the safety of the subjects, affect the efficacy evaluation or compliance, or other conditions that the researchers considered unsuitable for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Percentage (%) of body weight loss | Baseline to week 44
  Percentage (%) of body weight loss relative to baseline in both groups at week 44.

SECONDARY OUTCOMES:
Proportion of subjects with a body weight loss of ≥5% | Baseline to week 44
  Proportion of subjects with a body weight loss of ≥5% from baseline at week 44.
Waist circumference change from baseline | Baseline to week 44
  Waist circumference change from baseline at week 44.

CONTACTS AND LOCATIONS:
Locations (65):
- China (65):
  - Hefei Third People's Hospital, Hefei, Anhui
  - Xuancheng People'S Hospital, Xuancheng, Anhui
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Southwest Hospital of Amu, Chongqing, Chongqing Municipality
  - Fuling Hospital affiliated to Chongqing University, Chongqing, Chongqing Municipality
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Mengchao Hepatobiliary Hospital Of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Nanxishan Hospital of Guangxi Zhuang Autonomous Region, Guilin, Guangxi
  - Liuzhou People'S Hospital, Liuchow, Guangxi
  - The first Affiliated Hospital of GUANGXI medical university, Nanning, Guangxi
  - Wuzhou GongRen Hospital, Wuzhou, Guangxi
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - CangZhou Hospital of Integrated TCM-WM·HEBEI, Cangzhou, Hebei
  - The Affiliated Hospital of Chengde Medical College, Chengde, Hebei
  - Handan First Hospital, Handan, Hebei
  - Hebei Petro China Central Hospital, Langfang, Hebei
  - The Second Hospital Of Hebei Medical University, Shijiazhuang, Hebei
  - Tangshan GongRen Hospital, Tangshan, Hebei
  - Heilongjiang provincial hospital, Haerbin, Heilongjiang
  - The Third Affiliated Hospital of Qiqihar Medical College, Qiqihar, Heilongjiang
  - Anyang District Hospitai, Anyang, Henan
  - Luoyang Third People'S Hospital, Luoyang, Henan
  - The First affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - The Second Affiliated Hospital of Zhengzhou Univerisity, Zhengzhou, Henan
  - People'S Hospital of Zhengzhou, Zhengzhou, Henan
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - The Fourth Hospital of Changsha, Changsha, Hunan
  - Loudi Central Hospital, Loudi, Hunan
  - The Second People Hospital of Lianyungang, Lianyungang, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Jiangyin People' Hospital, Wuxi, Jiangsu
  - Jiangyin Hospital of Traditional Chinese Medicine, Wuxi, Jiangsu
  - XuZhou Cancer Hospital, Xuzhou, Jiangsu
  - XuZhou Central Hospital, Xuzhou, Jiangsu
  - First Affiliated Hospital Of Gannan Medical University, Ganzhou, Jiangxi
  - Xinyu People's Hospital, Xinyu, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Genertec Liaoyou Gem Flower Hospiital, Panjin, Liaoning
  - The sixth people's hospital at of Shenyang, Shenyang, Liaoning
  - Shanxi Provincial People's Hospital, Xi'an, Shaanxi
  - Xi'An International Medical Center Hospital, Xi'an, Shaanxi
  - Binzhou medical college affiliated hospital, Binzhou, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Affiliated Hospital of Jining Medical College, Jining, Shandong
  - Zibo Central Hospital, Zibo, Shandong
  - Shanghai Pudong New Area People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Jiading Central Hospital, Shanghai, Shanghai Municipality
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi, Shanxi
  - FIRST HOSPITAL OF SHANXI Medical, Taiyuan, Shanxi
  - The Affiliated Hospital of Southwet Medical University, Luzhou, Sichuan
  - Suining Central Hospital, Suining, Sichuan
  - The Second People's Hospital of Yibin City, Yibin, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Shihezi University, Shihezi, Xinjiang
  - The Second Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First People's Hospital of Xiaoshan District, Hangzhou, Zhejiang
  - Huzhou Center Hostipal, Huzhou, Zhejiang
  - Jiaxing Second Hospital, Jiaxing, Zhejiang
  - Ruian People's Hospital, Wenzhou, Zhejiang